CLINICAL TRIAL: NCT03355664
Title: A Multi-centre, Open-label Randomised Trial to Assess the Efficacy, Safety and Tolerability of the Triple ACT Artemether-lumefantrine+Amodiaquine (AL+AQ) Compared to the ACT Artemether-lumefantrine (AL) in Uncomplicated Falciparum Malaria in Cambodia and Vietnam
Brief Title: Study to Compare the Triple ACT AL+AQ With the ACT AL in Cambodia and Vietnam
Acronym: TACT-CV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAL17008
Record Dates: First submitted 2017-11-01; First posted 2017-11-28 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-03

CONDITIONS: Malaria, Falciparum
Keywords: Malaria, Falciparum; Malaria; Protozoan Infections; Lumefantrine; Artemether; Amodiaquine; Piperaquine; Artemether-lumefantrine combination; Artemisinins; Dihydroartemisinin; Mefloquine; Artemisinin; Antimalarials; Antiparasitic Agents; Anti-Infective Agents; ACT; TACT; Triple ACT(s); Resistance; Antimalarial resistance; Cardiotoxicity; Safety; Tolerability; Efficacy
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Protozoan Infections; Cardiotoxicity | interventions — bis(tetraheptylammonium)tetraiodocyclopentane tellurate(IV)

STUDY DESIGN:
Intervention Model Description: open-label randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT (Active Comparator): Artemether-lumefantrine for 3 days plus primaquine at hour 24
  Interventions: Drug: ACT
- TACT (Experimental): Artemether-lumefantrine for 3 days plus Amodiaquine for 3 days plus primaquine at hour 24
  Interventions: Drug: TACT

INTERVENTIONS:
Drug: ACT — Artemether-lumefantrine (20/120 mg) as a fixed dose combination twice daily for 3 days according to weight plus low dose primaquine at hour 24
  Arms: ACT
Drug: TACT — Artemether-lumefantrine (20/120 mg) as a fixed dose combination twice daily for 3 days according to weight plus Amodiaquine (150mg) twice daily for 3 days according to weight plus low dose primaquine at hour 24
  Arms: TACT

SUMMARY:
This study is a multi-centre, open-label randomised trial to assess the efficacy, safety and tolerability of the Triple ACT artemether-lumefantrine+amodiaquine (AL+AQ) compared to the ACT artemether-lumefantrine (AL) in uncomplicated falciparum malaria in Cambodia and Vietnam. The estimated total sample size is 600 patients from 2 sites in Cambodia and 2 sites in Vietnam. There are 2 treatment arms Arm 1: Artemether-lumefantrine for 3 days Arm 2: Artemether-lumefantrine for 3 days plus Amodiaquine for 3 days. According to the World Health Organization guideline, all patients except children under 10 kilograms will also be treated with a single dose of primaquine as a gametocytocidal treatment.

Funder :Bill & Melinda Gates Foundation (BMGF) Grant reference number: OPP1132628

DETAILED DESCRIPTION:
"The study of artemether-lumefantrine or artemether-lumefantrine combined with amodiaquine will be a two-arm randomized open label comparative study.

The main activity proposed is a series of detailed in vivo clinical, parasitological and pharmacological assessments in 600 subjects across 2 sites in Cambodian (400 subjects) and 2 sites in Vietnam (200 subjects). The subjects will be randomized between the ACT artemether-lumefantrine and the TACT artemether-lumefantrine+amodiaquine.

Parasite clearance rates will be assessed by repeated assessments of the parasite counts after the start of the antimalarial treatments. Efficacy, safety and tolerability of ACTs and TACTs will be assessed through weekly follow up visits where vital signs, symptom questionnaires, physical examinations, blood smears, biochemistry assays and full blood counts will be performed.

Ex vivo assessments of parasite susceptibility to artemisinins and partner drugs will be measured and compared to historical data, clinical phenotype and other sites in an effort to identify artemisinin and partner drug resistance.

This study will obtain data on the effect of antimalarials on the corrected QT intervals. In addition, the effects of antimalarials on factors such as post-treatment haematocrit and haemoglobin levels will be assessed. Extensive pharmacokinetic analysis will allow for an assessment of drug-drug interactions.

Plasma histidine-rich protein 2 (HRP2) levels (a marker of parasite biomass) that could potentially serve for the estimation of parasitaemia dynamics before and after treatment will be measured and subsequently modelled."

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 2 years to 65 years old
* Acute uncomplicated P. falciparum malaria, confirmed by positive blood smear with asexual forms of P. falciparum (or mixed with non-falciparum species)
* Asexual P. falciparum parasitaemia: 16 to 200,000/microlitre, determined on a thin or thick blood film
* Fever defined as > 37.5°C tympanic temperature or a history of fever within the last 24 hours
* Written informed consent (by parent/guardian in case of children)
* Willingness and ability of the patients or parents/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe/complicated malaria
* Haematocrit < 25% or Hb < 8 g/dL at screening
* Acute illness other than malaria requiring treatment
* For females: pregnancy, breast feeding
* Patients who have received artemisinin or a derivative or an artemisinin-containing combination therapy (ACT) within the previous 7 days
* History of allergy or known contraindication to artemisinins, lumefantrine or amodiaquine
* Previous splenectomy
* corrected QT interval > 450 milliseconds at moment of presentation
* Documented or claimed history of cardiac conduction problems
* Previous participation in the current study or another study in the previous 3 months

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Cambodia (2):
  - Siem Pang Health Center, Siem Pang, Stung Treng
  - Pailin Referral Hospital, Pailin
- Vietnam (2):
  - Hospital for Tropical Diseases of Khanh Hoa,, Vạn Giã, Khanh Hoa
  - Phuoc Long Hospital, Phước Long, Phuoc

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peto TJ, Tripura R, Callery JJ, Lek D, Nghia HDT, Nguon C, Thuong NTH, van der Pluijm RW, Dung NTP, Sokha M, Van Luong V, Long LT, Sovann Y, Duanguppama J, Waithira N, Hoglund RM, Chotsiri P, Chau NH, Ruecker A, Amaratunga C, Dhorda M, Miotto O, Maude RJ, Rekol H, Chotivanich K, Tarning J, von Seidlein L, Imwong M, Mukaka M, Day NPJ, Hien TT, White NJ, Dondorp AM. Triple therapy with artemether-lumefantrine plus amodiaquine versus artemether-lumefantrine alone for artemisinin-resistant, uncomplicated falciparum malaria: an open-label, randomised, multicentre trial. Lancet Infect Dis. 2022 Jun;22(6):867-878. doi: 10.1016/S1473-3099(21)00692-7. Epub 2022 Mar 8. PMID 35276064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled at hospitals and health centres 18 March 2018 to 30 January 2020
Pre-assignment Details: Actual number randomised was 312, however, an exclusion criterion was an ECG-measured QTc interval of ≥450ms. After randomisation the ECG was routinely repeated before drug administration, and in 2 participants (1 in each arm) the repeat ECG was ≥450 therefore no study drug was administered and the participants were treated with standard of care and recovered fully. There is no further data on these participants and the denominator for all subsequent tables is the 310 who received study drugs.
Groups:
- Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24: ACT: Artemether-lumefantrine (20/120 mg) as a fixed dose combination twice daily for 3 days according to weight plus low dose primaquine at hour 24
- Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24: TACT: Artemether-lumefantrine (20/120 mg) as a fixed dose combination twice daily for 3 days according to weight plus Amodiaquine (150mg) twice daily for 3 days according to weight plus low dose primaquine at hour 24
Period: Overall Study
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Started | 154 | 156
Completed | 139 | 144
Not Completed | 15 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 11 | 7
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24 | Total
Number analyzed (Participants) | 154 | 156 | 310
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [18 to 34] | 25 [19 to 33] | 25 [18 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 36
  Male | 142 | 132 | 274
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 25 | 26 | 51
  Cambodia | 129 | 130 | 259
Tympanic temperature ≥37·5°C [Count of Participants; unit: Participants] | 81 | 83 | 164
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 51 (11) | 51 (12) | 51 (12)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 158 (12) | 157 (14) | 158 (13)
Heart rate [Median (Inter-Quartile Range); unit: beats per minute (bpm)] | 89 [78 to 97] | 90 [81 to 104] | 90 [79 to 101]
Respiratory rate [Median (Inter-Quartile Range); unit: breaths per minute (bpm)] | 25 [23 to 28] | 26 [22 to 28] | 25 [22 to 28]
Systolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 113 (11) | 113 (12) | 113 (11)
Diastolic blood pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 69 (8) | 68 (8) | 69 (8)
Heart rate-corrected QT interval (QTcB) [Mean (Standard Deviation); unit: millisecond (ms)] | 413 (18) | 415 (17) | 414 (17)
Hemoglobin (Hb) [Mean (Standard Deviation); unit: grams per decilitre (g/dL)] | 12.8 (1.7) | 12.7 (1.8) | 12.7 (1.7)
Pfkelch13 mutant [Count of Participants; unit: Participants] | 81 | 93 | 174
Pfkelch13 wild-type [Count of Participants; unit: Participants] | 69 | 62 | 131
P. falciparum, not genotyped [Count of Participants; unit: Participants] | 4 | 1 | 5
Co-infection with P. vivax [Count of Participants; unit: Participants] | 22 | 29 | 51
Parasitaemia [Geometric Mean (Inter-Quartile Range); unit: Parasitaemias per µL] | 7670 [5356 to 10983] | 11647 [8538 to 15890] | 9464 [7467 to 11996]
Gametocytaemia [Count of Participants; unit: Participants] | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Polymerase Chain Reaction Corrected Efficacy Defined as Adequate Clinical and Parasitological Response (ACPR) by Study Arm
Description: Efficacy is defined as participants, following initial parasite and fever clearance, not having a recrudescence of the original plasmodium infection and fever, up to 42 days of follow up.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Participants | 146 | 151
Statistical Analysis 1: Comparison: Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 vs Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24; Test type: Superiority; p = 0.38, Regression, Cox; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.2 to 1.9]

2. Secondary Outcome: 42-day Polymerase Chain Reaction Corrected Efficacy According to Site/Geographic Region
Description: 42-day polymerase chain reaction corrected efficacy defined as adequate clinical and parasitological response (ACPR) according to site/geographic region.
Time Frame: 42 day
Population: The numbers analysed differ from the overall total as for this secondary analysis we report efficacy stratified by each of the 3 study sites.
Measure: Count of Participants; unit: Participants
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Participants
  West Cambodia: number analyzed (Participants) | 37 | 38
  West Cambodia | 32 | 35
  East Cambodia: number analyzed (Participants) | 92 | 92
  East Cambodia | 91 | 90
  Vietnam: number analyzed (Participants) | 25 | 26
  Vietnam | 23 | 26

3. Secondary Outcome: Parasite Clearance Half-life
Description: Parasite clearance half-life assessed by microscopy as primary parameter to determine parasite clearance
Time Frame: 42 day
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Hours | 5 (2.5) | 5.5 (2.6)

4. Secondary Outcome: Fever Clearance Time
Description: The time taken for the tympanic temperature to fall below 37.5˚C and remain there for at least 24 hours
Time Frame: 42 day
Measure: Mean (Standard Deviation); unit: Hours to fever clearance
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Hours to fever clearance | 18.3 (12.6) | 14.9 (9.9)

5. Secondary Outcome: Number of Severe Adverse Events by Study Arm
Description: All numerators in AE tables mean that the AE was reported as present according to the definitions defined in the US government DAIDS 2017 grading tables for reporting of adverse events. The AEs are reported without grading in this table, but are graded in the paper reporting this clinical trial.
  All Primary analyses are reported (also in the accepted manuscript) along with the secondary outcomes needed to support the primary analysis. Secondary outcomes not involving the randomised comparison will be updated when the analyses are available. Please note that analyses of these Secondary outcomes will take time.
Time Frame: 42 days
Measure: Number; unit: Participants
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Participants | 2 | 5

6. Secondary Outcome: Incidence of Adverse Events Concerning Markers of Hepatic or Renal Toxicity
Description: Total bilirubin, Alanine transaminase, Aspartate transaminase, Alkaline phosphatase and creatinine will be measured
Time Frame: 42 day
Measure: Number; unit: Events
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Events | 53 | 63

7. Secondary Outcome: Incidence of Prolongation of the Corrected QT Interval
Description: We record the number of events where the QT interval exceeds 500ms or increases by 60ms or greater.
Time Frame: 28 day
Measure: Number; unit: Events
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Events | 0 | 0

8. Secondary Outcome: Prolongation of the Corrected QT Interval
Description: We record the number of events where the QT interval exceeds 500ms or increases by 60ms or greater. There were zero events of this at any time point in either study arm. So no further analyses are possible.
Time Frame: Hour 4, Hour 24, Hour 28, Hour 48, Hour 52, Hour 60, Hour 64, Day 7 and Day 28 and between these time points
Measure: Number; unit: Events
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
Number analyzed (Participants) | 154 | 156
Events | 0 | 0

9. Secondary Outcome: Parasite Reduction Rates
Description: Parasite reduction rates and ratios at 24 and 48 hours assessed by microscopy
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 24 and 48 hours
Reporting Status: Not Posted, anticipated posting 2022-12

10. Secondary Outcome: Parasite Count to Fall 50%
Description: Time for parasite count to fall 50% of initial parasite density
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

11. Secondary Outcome: Parasite Count to Fall 90%
Description: Time for parasite count to fall 90% of initial parasite density
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

12. Secondary Outcome: Parasite Count to Fall 99%
Description: Time for parasite count to fall 99% of initial parasite density
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

13. Secondary Outcome: Change in Haematocrit
Description: Change in haematocrit at specified time points according to geographical location and study arm, stratified for G6PD status
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: Day 1 to 7, 14, 21, 28, 35, 42
Reporting Status: Not Posted, anticipated posting 2022-12

14. Secondary Outcome: Correlation Between the Host Genotype and the Pharmacokinetics and Pharmacodynamics of Antimalarials
Description: Correlation between the host genotype and the pharmacokinetics and pharmacodynamics of antimalarials
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 day
Reporting Status: Not Posted, anticipated posting 2022-12

15. Secondary Outcome: Proportion of Patients That Reports Completing a Full Course of Observed TACT or ACT
Description: Proportion of patients that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study because of drug related serious adverse event
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 day
Reporting Status: Not Posted, anticipated posting 2022-12

16. Secondary Outcome: Prevalence of Kelch13 Mutations of Known Significance
Description: Prevalence of Kelch13 mutations of known significance
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 day
Reporting Status: Not Posted, anticipated posting 2022-12

17. Secondary Outcome: Prevalence/Incidence of Other Genetic Markers of Antimalarial Drug Resistance Such as Multidrug Resistance Gene 1 Copy Number and Multidrug Resistance Gene 1 Mutations
Description: Prevalence/incidence of other genetic markers of antimalarial drug resistance such as multidrug resistance gene 1 copy number and multidrug resistance gene 1 mutations
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 48 hours
Reporting Status: Not Posted, anticipated posting 2022-12

18. Secondary Outcome: Genome Wide Association With in Vivo/in Vitro Sensitivity Parasite Phenotype
Description: Genome wide association with in vivo/in vitro sensitivity parasite phenotype
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 day
Reporting Status: Not Posted, anticipated posting 2022-12

19. Secondary Outcome: Correlation Between Single Nucleotide Polymorphisms and Whole Genome Sequencing
Description: Correlation between single nucleotide polymorphisms measured in dry blood spots and whole genome sequencing in leukocyte depleted blood samples
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 day
Reporting Status: Not Posted, anticipated posting 2022-12

20. Secondary Outcome: A Comparison of Transcriptomic Patterns Between Sensitive and Resistant Parasites
Description: Transcriptomic patterns measure at baseline and at specified time points after the start of treatment comparing sensitive and resistant parasites.
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: baseline and t = 6 hours
Reporting Status: Not Posted, anticipated posting 2022-12

21. Secondary Outcome: Correlation Between Quantitative Polymerase Chain Reaction Based Versus Microscopy Based Assessments of Parasite Clearance Dynamics
Description: Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2022-12

22. Secondary Outcome: Proportion of Patients With Gametocytaemia Before, During and After Treatment With TACT or ACT
Description: Proportion of patients with gametocytaemia before, during and after treatment with TACT or ACT stratified by the presence of gametocytes at enrolment
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: At admission and up to day 14
Reporting Status: Not Posted, anticipated posting 2022-12

23. Secondary Outcome: Levels of RNA Transcription Coding for Male or Female Specific Gametocytes
Description: Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2022-12

24. Secondary Outcome: In Vitro Sensitivity of P. Falciparum to Artemisinins and Partner Drugs
Description: In vitro sensitivity of P. falciparum to artemisinins and partner drugs according to study sites and genotype
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: At admission & subjects with recurrent parasitaemia, up to 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

25. Secondary Outcome: Pharmacokinetic Profiles and Interactions (Cmax) of Artemisinin-derivatives and Partner Drugs
Description: Pharmacokinetic profiles and interactions (Cmax) of artemisinin-derivatives and partner drugs in 20 ACT treated and 20 TACT treated patients of both study arms in Vietnam
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

26. Secondary Outcome: Pharmacokinetic Profiles and Interactions (AUC) of Artemisinin-derivatives and Partner Drugs
Description: Pharmacokinetic profiles and interactions (AUC) of artemisinin-derivatives and partner drugs in 20 ACT treated and 20 TACT treated patients of both study arms in Vietnam
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

27. Secondary Outcome: Day 7 Drug Levels of Partner Drugs in Association With Treatment Efficacy and Treatment Arm
Description: Day 7 drug levels of partner drugs in association with treatment efficacy and treatment arm
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 7 days
Reporting Status: Not Posted, anticipated posting 2022-12

28. Secondary Outcome: Correlation Between Histidine-rich Protein 2 (HRP2) Based Versus Microscopy Based Assessments of Parasite Clearance Dynamics
Description: Correlation between histidine-rich protein 2 (HRP2) based versus microscopy based assessments of parasite clearance dynamics
  The data are collected, but this secondary outcome will come from analyses done by specialist researchers and the results will not affect the the presently reported primary outcomes of efficacy, safety and tolerability. These fields will be updated once results become available. We will also provide a link to the paper reporting the trial when it is published online as this will provide additional detail about the study.
Time Frame: 42 days
Reporting Status: Not Posted, anticipated posting 2022-12

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/156
Serious Adverse Events (participants affected / at risk) | 2/154 | 5/156
Other Adverse Events (participants affected / at risk) | 122/154 | 141/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 (N=154) | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24 (N=156)
gastritis (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
severe malaria (Infections and infestations) | 0 | 2
dengue (Infections and infestations) | 1 | 0
Transaminitis (Hepatobiliary disorders) | 0 | 1
anaemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artemether-lumefantrine for 3 Days Plus Primaquine at Hour 24 (N=154) | Artemether-lumefantrine for 3 Days Plus Amodiaquine for 3 Days Plus Primaquine at Hour 24 (N=156)
vomiting (Gastrointestinal disorders) | 3 | 12
nausea (Gastrointestinal disorders) | 3 | 11
dizziness (General disorders) | 9 | 16
abdominal pain (Gastrointestinal disorders) | 19 | 22
diarrhoea (Gastrointestinal disorders) | 13 | 17
headache (General disorders) | 19 | 20
fatigue (General disorders) | 11 | 15
loss of appetite (General disorders) | 9 | 9
itching (Skin and subcutaneous tissue disorders) | 2 | 5
blurred vision (Eye disorders) | 7 | 4
sleep disturbance (General disorders) | 8 | 12
suicidal ideation (Psychiatric disorders) | 0 | 0
pyschiatric problems (Psychiatric disorders) | 0 | 0
creatinine (Renal and urinary disorders) | 4 | 10
total bilirubin (Hepatobiliary disorders) | 2 | 0
alkaline phosphatase (ALP) (Hepatobiliary disorders) | 14 | 8
alanyl transferase (ALT) (Hepatobiliary disorders) | 16 | 21
aspartate transferase (AST) (Hepatobiliary disorders) | 17 | 24
anaemia (Blood and lymphatic system disorders) | 27 | 46
leukocytopenia (Blood and lymphatic system disorders) | 2 | 0
neutropenia (Blood and lymphatic system disorders) | 1 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 38 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03355664/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT03355664/SAP_001.pdf